CLINICAL TRIAL: NCT00359632
Title: Prospective Study Of Ophthalmologic Function In Patients Receiving Linezolid For Six Weeks Or Greater
Brief Title: Study to Evaluate Eye Function in Patients Taking Linezolid for Six Weeks or Greater
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped due to poor enrollment on 28 Feb 2012. Reason for termination was not due to safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: A5951110; 2006-002303-14 (EudraCT Number)
Record Dates: First submitted 2006-07-28; First posted 2006-08-02 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Optic Nerve Diseases
Keywords: Optic neuropathy following long-term linezolid use
MeSH Terms: conditions — Optic Nerve Diseases | interventions — Case-Control Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linezolid (Experimental): Subjects have received at least 6 weeks of linezolid therapy (600 mg BID). Continued duration of linezolid treatment is based on treating physician's benefit/risk assessment. A matching control who did not receive linezolid will be selected for each linezolid treated subject.
  Interventions: Drug: Zyvox - linezolid
- Matched control (Active Comparator): Control subjects individually matched to linezolid subjects (on age, gender and type of infection) who received at least 6 weeks of antibiotics other than linezolid. Control group assessed only at baseline visit to assess presence of background abnormalities in the study test panel.
  Interventions: Drug: Matched control

INTERVENTIONS:
Drug: Zyvox - linezolid — Observation and testing in patients for whom their treating physician has determined linezolid is an appropriate therapy. Eye tests performed for subjects who have received linezolid for at least 6 weeks and matching controls who have received other antibiotics for similar types of infections.
  Arms: Linezolid
Drug: Matched control — Matched controls received an antibiotic other than linezolid for at least 6 weeks prior to baseline visit. The control group had only a baseline visit and there were no post baseline study visits.
  Arms: Matched control

SUMMARY:
To understand and characterize the effects of linezolid on the optic nerve by observing and following patients who have been treated with linezolid for six weeks or longer for the development of signs or symptoms of visual disturbance or eye disorders.

DETAILED DESCRIPTION:
Characterize Optic Side Effect

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who are 18 years of age or older.
* Subjects in Treated Group:
* Subjects must have received linezolid 600 mg BID for six weeks or greater and be currently on drug (or have received linezolid within 7 days of baseline evaluation).
* Subjects who have current signs or symptoms compatible with linezolid toxicity (i.e. optic or peripheral neuropathy) may be enrolled in the study if they are on linezolid at time of baseline evaluation (or have received linezolid within 7 days of baseline evaluation).
* Linezolid may be discontinued at any time at the primary physician's discretion and remain on the study.
* Women of childbearing potential must use adequate contraception
* Subjects in Control Group:
* Subjects will have a diagnosis similar to patients in the treated group and similar important co-morbidities and epidemiologic factors if possible.

Exclusion Criteria:

* Subject in Treated Group:
* Subjects with a known presence of optic or peripheral nerve damage due to another illness, condition or medication.
* Subjects with a pre-existing or a diagnosis at time of screening visit of an ophthalmologic condition that would adversely affect the study testing protocol (e.g. dense cataracts, macular degeneration, retinitis pigmentosa).
* Subjects who are currently receiving or anticipated to receive another medication, antibiotic or other, that has known potential to produce ocular or neurologic toxicity indistinguishable from that caused by linezolid or lactic acidosis.
* Subjects with a history of significant exposure, in the opinion of the investigator and with prior discussion with the medical monitor, to medications known to produce optic or peripheral neuropathy.
* Subjects with an active communicable disease (i.e., tuberculosis assessed as currently communicable) and subjects on active treatment for tuberculosis or other mycobacterial disease that include drugs that have known potential to produce ocular or neurologic toxicity.
* Subjects with severe liver disease or abnormal liver function test.
* Subjects in Control Group:
* Subjects must not currently be taking linezolid or have received it for more than 7 days at any time.
* Subjects with a known presence of optic or peripheral nerve damage due to another illness, condition or medication.
* Subjects with a pre-existing or a diagnosis at the screening visit of an ophthalmologic condition that would adversely affect the study testing protocol (e.g. dense cataracts, macular degeneration, retinitis pigmentosa).
* Subjects who are currently receiving another medication, antibiotic or other, that has known potential to produce ocular or neurologic toxicity indistinguishable from that caused by linezolid or lactic acidosis.
* Subjects with a history of significant exposure, in the opinion of the investigator and with prior discussion with the medical monitor, to medications known to produce optic or peripheral neuropathy.
* Subjects with an active communicable disease (i.e., tuberculosis assessed as currently communicable) and subjects on active treatment for tuberculosis or other mycobacterial disease that include drugs that have known potential to produce ocular or neurologic toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (7):
  - St. Bernards Research Center, Jonesboro, Arkansas
  - Triple O Research Institute, PA, West Palm Beach, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Department of Medicine/Division of Infectious Diseases, Minneapolis, Minnesota
  - Drexel University College of Medicine, Partnership Comprehensive Care Practice, Philadelphia, Pennsylvania
  - Associates in Infectious Disease and Tropical Medicine, Pittsburgh, Pennsylvania
- Italy (4):
  - Azienda Ospedaliera Universitaria di San Martino, Genova
  - Ospedale San Martino, Clinica Malattie Infettive, Genova
  - Università di Genova, Genova
  - Clinica Malattie Infettive, Azienda Ospedaliero Universitaria Santa Maria della Misericordia, Udine
- Infektionskliniken 1-73, Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951110&StudyName=Study%20to%20Evaluate%20Eye%20Function%20in%20Patients%20Taking%20Linezolid%20for%20Six%20Weeks%20or%20Greater

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine centers (2 centers in Italy, 1 center in Sweden, and 6 centers in the US) enrolled subjects for inclusion in the study. Sites were selected based on their capability to perform the comprehensive testing and to treat types of infections that might require therapy with linezolid for 6 weeks or longer.
Pre-assignment Details: There were separate selection criteria for subjects in the treated and control groups. At the Screening/Baseline visit (Day 1), subjects were eligible for the study after verification that they met the relevant inclusion/exclusion criteria and the study had been explained to them.
Groups:
- Linezolid: Participants received linezolid either as tablets, by mouth (PO) or as an intravenous (IV) infusion at a dose of 600 milligrams (mg), twice daily (BID). Mode of administration and duration of treatment was at the discretion of the investigator, but for study purposes, the participant had to receive linezolid treatment for a minimum of 6 weeks (at least 42 days).
- Control: Control participants individually matched to linezolid participants (on age, gender, and type of infection) received antibiotics other than linezolid per standard of care at the discretion of the treating investigator, for at least 6 weeks (at least 42 days). The control group was only assessed at the baseline visit to identify the presence of background abnormalities in the study test panel.
Period: Overall Study
Arm/Group | Linezolid | Control
Started | 24 | 9
Completed | 20 | 9
Not Completed | 4 | 0
Not completed — Death | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance with visit schedule | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Linezolid: Participants received linezolid either as tablets, PO or as an IV infusion at a dose of 600 mg, BID. Mode of administration and duration of treatment was at the discretion of the investigator, but for study purposes, the participant had to receive linezolid treatment for a minimum of 6 weeks (at least 42 days).
- Total: Total of all reporting groups
Arm/Group | Linezolid | Control | Total
Number analyzed (Participants) | 24 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (13.38) | 50.1 (11.86) | 52.5 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 14 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event
Time Frame: Through and including 28 calendar days after the last administration of the investigational product
Measure: Number; unit: Percentage of Participants
Arm/Group | Linezolid | Control
Number analyzed (Participants) | 24 | 9
Percentage of Participants
  Adverse events, % | 83.3 | 11.1
  Serious adverse events, % | 25.0 | 0
  Severe adverse events, % | 12.5 | 0
  Discontinued due to adverse events, % | 29.2 | 0
  Dose Reduced or Temporary Discontinuation, % | 12.5 | 0

2. Secondary Outcome: Percentage of Participants by Clinical Outcome of Infection at End of Study
Description: Clinical response was evaluated at the End of Study visit (30 days after last dose) as Cure, Improvement, Failure, Unknown or Other. Clinical response was based primarily on the global assessment of the clinical presentation of the subject made by the investigator at that evaluation timepoint. The clinical response classifications were defined as follows. Cure: Resolution of the clinical signs and symptoms of infection, when compared to Baseline. No additional antimicrobial treatment is required for the disease under study. Improvement: Improvement in 2 or more, but not all, of the clinical signs and symptoms of infection, when compared with Baseline. No additional antimicrobial treatment is required for the disease under study. Failure: Persistence or progression of Baseline clinical signs and symptoms of infection, or development of new clinical findings consistent with active infection. Unknown: Inability to assess clinical response.
Time Frame: At End of Study visit
Measure: Number; unit: Percentage of Participants
Arm/Group | Linezolid
Number analyzed (Participants) | 21
Percentage of Participants
  Cure, % | 47.6
  Improvement, % | 42.9
  Failure, % | 0
  Unknown, % | 0
  Other, % | 9.5

ADVERSE EVENTS:
Time Frame: Through and including 28 calendar days after the last administration of the investigational product
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid | Control
Serious Adverse Events (participants affected / at risk) | 6/24 | 0/9
Other Adverse Events (participants affected / at risk) | 20/24 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linezolid (N=24) | Control (N=9)
Erythropoiesis abnormal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sideroblastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Linezolid (N=24) | Control (N=9)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 1 (1) | 0 (0)
Narrow anterior chamber angle (Eye disorders) | 0 (0) | 1 (1)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal disorder (Eye disorders) | 1 (1) | 0 (0)
Toxic optic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0/1 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Tooth discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 2 (2) | 0 (0)
Protein total increased (Investigations) | 1 (1) | 0 (0)
Vitamin B1 decreased (Investigations) | 1 (1) | 0 (0)
Vitamin B12 decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Vitamin B6 deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This pilot study was exploratory and not designed to be powered for safety or efficacy. Controls were not followed post-baseline whereas linezolid patients returned for multiple study visits. The study was terminated early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No